CLINICAL TRIAL: NCT02189200
Title: Effect of Nutritional Counseling Associated With the Ingestion of Oat Bran in Hypercholesterolemic Subjects in Secondary Prevention
Brief Title: Nutritional Counseling Associated With the Ingestion of Oat Bran in Hypercholesterolemic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Simone Raimondi de Souza, Dra., Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03131712.3.0000.5265
Record Dates: First submitted 2014-07-07; First posted 2014-07-14 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Dietary Modification
Keywords: nutritional counseling; oat bran; dyslipidemia; cardiovascular disease
MeSH Terms: conditions — Dyslipidemias; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oat bran group (Active Comparator): oat bran (40g per day)
  Interventions: Dietary Supplement: oat bran - 40g
- Placebo group (Placebo Comparator): refined rice flour (40g per day)
  Interventions: Dietary Supplement: refined rice flour- 40g

INTERVENTIONS:
Dietary Supplement: oat bran - 40g — oat bran - 40g per day
  Arms: Oat bran group
Dietary Supplement: refined rice flour- 40g — refined rice flour - 40g per day
  Arms: Placebo group

SUMMARY:
Dyslipidemia is among the risk factors for cardiovascular diseases (CVD). Is's due to genetic and / or environmental factors such as inadequate dietary pattern. The occurrence of adverse events with statins, added to recent questions about their benefits on hard outcomes, opens a gap for the importance of seeking other forms of treatment of dyslipidemia, particularly in patients for secondary prevention. The consumption of oat bran, beta-glucan source of dietary fibers with supposed action in reducing the absorption of exogenous cholesterol and the endogenous synthesis of it, and source of avenanthramides, phytochemical compounds with alleged antioxidant in lipid membranes, can be effective strategy for secondary prevention of atherosclerotic disease.

DETAILED DESCRIPTION:
Objectives: To evaluate the effect of nutritional counseling associated with the consumption of oat bran (40g per day) in lowering cholesterol, glucose profile and anthropometric parameters of subjects in secondary prevention, evaluate the quality of the diet and the intake of processed foods and ingredients added.

Methods: A randomized block, double-blind, placebo-controlled trial lasting 90 days. Inclusion criteria: individuals aged greater than 20 years, both genders, with LDL-c equal or higher than 130mg/dL fasting lipemia. Eligible individuals were considered using oral lipid-lowering, since the dose reported in the early nutritional intervention was maintained during the study. Exclusion criteria: patients requiring reduction in daily fluid intake, supplement use in dietary fiber and gestation / lactation. Data collected: gender; age; education; drugs; body mass (BM), height, body mass index (BMI), waist circumference (WC), neck circumference (NC); blood pressure; dietary surveys, total cholesterol (TC), LDL-C, HDL-cholesterol (HDL-c), triglycerides (TG), fasting glucose (GLU), fasting insulin (INS), HOMA-IR and QUICK. The diet quality was evaluated at baseline and end of study through the Diet Quality Index Revised (IQD-R). The sample size calculation was performed from a pilot study. It came to the need for 63 subjects for each group, oat bran group (GFAV) and placebo group (GPL). The level of statistical significance was 5% (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* LDL-c equal or higher than 130mg/dL fasting lipemia.

Exclusion Criteria:

* patients requiring reduction in daily fluid intake
* patients in use of dietary fiber supplements
* gestation
* lactation

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in LDL-cholesterol in three months | mesures assessed in baseline, after 30, 60 and 90 days

SECONDARY OUTCOMES:
Change from baseline in glucose profile in three months | mesures assessed in baseline, after 30, 60 and 90 days

OTHER OUTCOMES:
Change from baseline in body mass | mesures in kg, assessed in baseline, after 30, 60 and 90 days
Change from baseline in waist circumference | mesures in cm, assessed in baseline, after 30, 60 and 90 days
Change from baseline in neck circumference | mesures in cm, assessed in baseline, after 30, 60 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Simone R. Souza, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Instituto Estadual de Cardiologia Aloysio de Castro - IECAC, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Adamsson V, Reumark A, Marklund M, Larsson A, Riserus U. Role of a prudent breakfast in improving cardiometabolic risk factors in subjects with hypercholesterolemia: a randomized controlled trial. Clin Nutr. 2015 Feb;34(1):20-6. doi: 10.1016/j.clnu.2014.04.009. Epub 2014 Apr 21. PMID 24814382
- [Background] Andersson KE, Hellstrand P. Dietary oats and modulation of atherogenic pathways. Mol Nutr Food Res. 2012 Jul;56(7):1003-13. doi: 10.1002/mnfr.201100706. Epub 2012 Jun 12. PMID 22764134
- [Background] Bentzon JF, Otsuka F, Virmani R, Falk E. Mechanisms of plaque formation and rupture. Circ Res. 2014 Jun 6;114(12):1852-66. doi: 10.1161/CIRCRESAHA.114.302721. PMID 24902970
- [Background] Briel M, Vale N, Schwartz GG, de Lemos JA, Colivicchi F, den Hartog FR, Ostadal P, Macin SM, Liem A, Mills E, Bhatnagar N, Bucher HC, Nordmann AJ. Updated evidence on early statin therapy for acute coronary syndromes: meta-analysis of 18 randomized trials involving over 14,000 patients. Int J Cardiol. 2012 Jun 28;158(1):93-100. doi: 10.1016/j.ijcard.2011.01.033. Epub 2011 Feb 4. PMID 21295870
- [Background] Sadiq Butt M, Tahir-Nadeem M, Khan MK, Shabir R, Butt MS. Oat: unique among the cereals. Eur J Nutr. 2008 Mar;47(2):68-79. doi: 10.1007/s00394-008-0698-7. Epub 2008 Feb 26. PMID 18301937
- [Background] Camargo A, Meneses ME, Perez-Martinez P, Delgado-Lista J, Jimenez-Gomez Y, Cruz-Teno C, Tinahones FJ, Paniagua JA, Perez-Jimenez F, Roche HM, Malagon MM, Lopez-Miranda J. Dietary fat differentially influences the lipids storage on the adipose tissue in metabolic syndrome patients. Eur J Nutr. 2014;53(2):617-26. doi: 10.1007/s00394-013-0570-2. Epub 2013 Aug 7. PMID 23922010
- [Background] Charlton KE, Tapsell LC, Batterham MJ, O'Shea J, Thorne R, Beck E, Tosh SM. Effect of 6 weeks' consumption of beta-glucan-rich oat products on cholesterol levels in mildly hypercholesterolaemic overweight adults. Br J Nutr. 2012 Apr;107(7):1037-47. doi: 10.1017/S0007114511003850. Epub 2011 Aug 3. PMID 21810288
- [Background] Chen CY, Milbury PE, Kwak HK, Collins FW, Samuel P, Blumberg JB. Avenanthramides and phenolic acids from oats are bioavailable and act synergistically with vitamin C to enhance hamster and human LDL resistance to oxidation. J Nutr. 2004 Jun;134(6):1459-66. doi: 10.1093/jn/134.6.1459. PMID 15173412
- [Background] Guo W, Wise ML, Collins FW, Meydani M. Avenanthramides, polyphenols from oats, inhibit IL-1beta-induced NF-kappaB activation in endothelial cells. Free Radic Biol Med. 2008 Feb 1;44(3):415-29. doi: 10.1016/j.freeradbiomed.2007.10.036. Epub 2007 Oct 22. PMID 18062932
- [Background] Handelman GJ, Cao G, Walter MF, Nightingale ZD, Paul GL, Prior RL, Blumberg JB. Antioxidant capacity of oat (Avena sativa L.) extracts. 1. Inhibition of low-density lipoprotein oxidation and oxygen radical absorbance capacity. J Agric Food Chem. 1999 Dec;47(12):4888-93. doi: 10.1021/jf990529j. PMID 10606548
- [Background] Jenkins DJ, Kendall CW, Vuksan V, Vidgen E, Parker T, Faulkner D, Mehling CC, Garsetti M, Testolin G, Cunnane SC, Ryan MA, Corey PN. Soluble fiber intake at a dose approved by the US Food and Drug Administration for a claim of health benefits: serum lipid risk factors for cardiovascular disease assessed in a randomized controlled crossover trial. Am J Clin Nutr. 2002 May;75(5):834-9. doi: 10.1093/ajcn/75.5.834. PMID 11976156
- [Background] Jenkins AL, Jenkins DJ, Wolever TM, Rogovik AL, Jovanovski E, Bozikov V, Rahelic D, Vuksan V. Comparable postprandial glucose reductions with viscous fiber blend enriched biscuits in healthy subjects and patients with diabetes mellitus: acute randomized controlled clinical trial. Croat Med J. 2008 Dec;49(6):772-82. doi: 10.3325/cmj.2008.49.722. PMID 19090602
- [Background] Jenkins DJ, Jones PJ, Lamarche B, Kendall CW, Faulkner D, Cermakova L, Gigleux I, Ramprasath V, de Souza R, Ireland C, Patel D, Srichaikul K, Abdulnour S, Bashyam B, Collier C, Hoshizaki S, Josse RG, Leiter LA, Connelly PW, Frohlich J. Effect of a dietary portfolio of cholesterol-lowering foods given at 2 levels of intensity of dietary advice on serum lipids in hyperlipidemia: a randomized controlled trial. JAMA. 2011 Aug 24;306(8):831-9. doi: 10.1001/jama.2011.1202. PMID 21862744
- [Background] Kaestner R, Darden M, Lakdawalla D. Are investments in disease prevention complements? The case of statins and health behaviors. J Health Econ. 2014 Jul;36:151-63. doi: 10.1016/j.jhealeco.2014.04.006. Epub 2014 Apr 16. PMID 24814322
- [Background] Kalantarian S, Rimm EB, Herrington DM, Mozaffarian D. Dietary macronutrients, genetic variation, and progression of coronary atherosclerosis among women. Am Heart J. 2014 Apr;167(4):627-635.e1. doi: 10.1016/j.ahj.2014.01.001. Epub 2014 Jan 15. PMID 24655714
- [Background] Keaney JF Jr. Immune modulation of atherosclerosis. Circulation. 2011 Nov 29;124(22):e559-60. doi: 10.1161/CIRCULATIONAHA.111.074096. No abstract available. PMID 22125193
- [Background] Lee DS, Markwardt S, Goeres L, Lee CG, Eckstrom E, Williams C, Fu R, Orwoll E, Cawthon PM, Stefanick ML, Mackey D, Bauer DC, Nielson CM. Statins and physical activity in older men: the osteoporotic fractures in men study. JAMA Intern Med. 2014 Aug;174(8):1263-70. doi: 10.1001/jamainternmed.2014.2266. PMID 24911216
- [Background] Maki KC, Beiseigel JM, Jonnalagadda SS, Gugger CK, Reeves MS, Farmer MV, Kaden VN, Rains TM. Whole-grain ready-to-eat oat cereal, as part of a dietary program for weight loss, reduces low-density lipoprotein cholesterol in adults with overweight and obesity more than a dietary program including low-fiber control foods. J Am Diet Assoc. 2010 Feb;110(2):205-14. doi: 10.1016/j.jada.2009.10.037. PMID 20102847
- [Background] Moodie R, Stuckler D, Monteiro C, Sheron N, Neal B, Thamarangsi T, Lincoln P, Casswell S; Lancet NCD Action Group. Profits and pandemics: prevention of harmful effects of tobacco, alcohol, and ultra-processed food and drink industries. Lancet. 2013 Feb 23;381(9867):670-9. doi: 10.1016/S0140-6736(12)62089-3. Epub 2013 Feb 12. PMID 23410611
- [Background] Nie L, Wise ML, Peterson DM, Meydani M. Avenanthramide, a polyphenol from oats, inhibits vascular smooth muscle cell proliferation and enhances nitric oxide production. Atherosclerosis. 2006 Jun;186(2):260-6. doi: 10.1016/j.atherosclerosis.2005.07.027. Epub 2005 Sep 1. PMID 16139284
- [Background] Rojas-Fernandez CH, Goldstein LB, Levey AI, Taylor BA, Bittner V, The National Lipid Association's Safety Task Force. An assessment by the Statin Cognitive Safety Task Force: 2014 update. J Clin Lipidol. 2014 May-Jun;8(3 Suppl):S5-16. doi: 10.1016/j.jacl.2014.02.013. PMID 24793442
- [Background] Smith SC Jr, Benjamin EJ, Bonow RO, Braun LT, Creager MA, Franklin BA, Gibbons RJ, Grundy SM, Hiratzka LF, Jones DW, Lloyd-Jones DM, Minissian M, Mosca L, Peterson ED, Sacco RL, Spertus J, Stein JH, Taubert KA. AHA/ACCF secondary prevention and risk reduction therapy for patients with coronary and other atherosclerotic vascular disease: 2011 update: a guideline from the American Heart Association and American College of Cardiology Foundation endorsed by the World Heart Federation and the Preventive Cardiovascular Nurses Association. J Am Coll Cardiol. 2011 Nov 29;58(23):2432-46. doi: 10.1016/j.jacc.2011.10.824. Epub 2011 Nov 3. No abstract available. PMID 22055990
- [Background] Wolever TM, Gibbs AL, Brand-Miller J, Duncan AM, Hart V, Lamarche B, Tosh SM, Duss R. Bioactive oat beta-glucan reduces LDL cholesterol in Caucasians and non-Caucasians. Nutr J. 2011 Nov 25;10:130. doi: 10.1186/1475-2891-10-130. PMID 22118569
- [Background] Yang J, Ou B, Wise ML, Chu Y. In vitro total antioxidant capacity and anti-inflammatory activity of three common oat-derived avenanthramides. Food Chem. 2014 Oct 1;160:338-45. doi: 10.1016/j.foodchem.2014.03.059. Epub 2014 Mar 21. PMID 24799247
- [Background] Zhang J, Li L, Song P, Wang C, Man Q, Meng L, Cai J, Kurilich A. Randomized controlled trial of oatmeal consumption versus noodle consumption on blood lipids of urban Chinese adults with hypercholesterolemia. Nutr J. 2012 Aug 6;11:54. doi: 10.1186/1475-2891-11-54. PMID 22866937
- See also: WORLD HEALTH ORGANIZATION. Cardiovascular disease prevention and control. Translating evidence into action, 2005 — http://apps.who.int/iris/bitstream/10665/43235/1/9241593253_eng.pdf?ua=1
- See also: WORLD HEALTH ORGANIZATION. Prevention of cardiovascular disease: guidelines for assessment and management of total cardiovascular risk, 2007 — http://whqlibdoc.who.int/publications/2007/9789241547178_eng.pdf?ua=1